CLINICAL TRIAL: NCT04097301
Title: A Phase I-IIa Trial to Assess the Safety and Antitumor Activity of Autologous CD44v6 CAR T-cells in Acute Myeloid Leukemia and Multiple Myeloma Expressing CD44v6
Brief Title: Study of CAR T-cell Therapy in Acute Myeloid Leukemia and Multiple Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Inability to close the study in a clinically relevant time frame
Sponsor: AGC Biologics S.p.A. (Industry)
Collaborators: Horizon 2020 - European Commission (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EURE-CART-1; 2018-000813-19 (EudraCT Number)
Record Dates: First submitted 2019-08-05; First posted 2019-09-20 (Actual); Results first posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2021-12

CONDITIONS: Acute Myeloid Leukemia; Multiple Myeloma
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Multiple Myeloma | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MLM-CAR44.1 T-cells infusion (Experimental): PHASE I: i.v. single dose of MLM-CAR44.1 T-cells: 0.5 x 10E6/Kg or 1 x 10E6/Kg or 2 x10E6/Kg according to the BOIN design.
  PHASE IIa: i.v. single dose of MLM-CAR44.1 T-cells corresponding to the maximum tolerated dose (MTD).
  Phase I and IIa Pre-treatment: lymphodepleting chemotherapy with cyclophosphamide (500 mg/m2) and fludarabine (30 mg/m2) daily from day -5 to day -3
  Interventions: Drug: MLM-CAR44.1 T-cells at day 0 Single intravenous infusion

INTERVENTIONS:
Drug: MLM-CAR44.1 T-cells at day 0 Single intravenous infusion — Lymphodepleting chemotherapy with cyclophosphamide (500 mg/m2) and fludarabine (30 mg/m2) daily from day -5 to day -3.
  Other Names: CAR-T cells

SUMMARY:
The purpose of this first-in-man Phase I-IIa study is to evaluate the safety and antitumor activity of autologous CD44v6 CAR T-cells in patients with acute myeloid leukemia (AML) and multiple myeloma (MM).

DETAILED DESCRIPTION:
The study is a seamless Phase I/IIa, open-label, multicenter clinical trial that combines Phase I dose escalation based on toxicity with Phase IIa dose expansion based on antitumor activity. Considering the "first in human" nature of this clinical study, the Bayesian Optimal Interval Design (BOIN) has been chosen to minimize any risks of exposure to the novel CD44v6 CAR T-cells during dose escalation. The study population is made up of patients with relapsed/refractory AML or MM expressing CD44v6.

The medicinal product under investigation (MLM-CAR44.1 T-cells) is patient specific as it is prepared starting from lymphocytes of the patient collected through lymphocyte apheresis. These autologous T-cells are expanded in vitro in large numbers and genetically modified to express the CAR CD44v6ΔNL gene and thus acquire antitumor functions. As a safety feature, the MLM-CAR44.1 T-cells are genetically modified to also express the HSV-TK Mut2 gene (suicide gene), which can be selectively activated in case of severe toxicity through the administration of ganciclovir (GCV), leading to the death of proliferating CAR T-cells.

The aim of this study is to assess the safety, antitumor activity and feasibility of CD44v6 CAR T cell immunotherapy in AML and MM.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all the following inclusion criteria to be eligible for the study.

1. Written informed consent before any study-related procedure.
2. Adults and children:

   1. Adults 18 to 75 (65) years old with AML or MM.
   2. Children 1 to 17 years old with AML, only in Phase IIa.
3. Confirmed diagnosis of AML or MM as follows:

   1. AML: Primary or secondary AML (any subtype except acute promyelocytic leukemia) according to World Health Organization (WHO) classification.
   2. MM with measurable disease as defined by the International Myeloma Working Group (IMWG).
4. Patients with relapse or refractory disease:

   1. AML patients must be unlikely to benefit from cytotoxic chemotherapy as follows:

      * Leukemia refractory to at least 2 induction attempts.
      * Leukemia in relapse within 1 year following complete response (CR) after at least 2 induction attempts.
      * High-risk leukemia in adults according to 2017 European LeukemiaNet (ELN) in first relapse after a hypomethylating agent or a cycle containing cytarabine at a dose ≥ 1g/sqm a day (e.g. FLAG-IDA), except for FLT3-mutated AML.
      * High-risk leukemia in children as defined by the Italian Association of Pediatric Hematology and Oncology (AIEOP).
   2. Patients with MM must have a relapse or refractory disease after at least 4 different prior treatments in 3 treatment lines, or 4 treatments in 2 treatment lines in case of early relapsing patients (relapse in less than 1.5 years). Treatments include:

      * Proteasome inhibitor
      * High-dose alkylating agent if patients less than 70 years old
      * Immunomodulatory drug (IMID)
      * A monoclonal antibody (i.e. anti CD38 monoclonal antibody)
5. Positive CD44v6 expression on tumor cells by flow cytometry.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
7. Life expectancy of at least 12 weeks.
8. Adequate organ function (hepatic, cardiac, pulmonary).
9. Recovery from toxicities of clinical consequence attributed to previous chemotherapy to CTCAE v5.0 Grade 1 (i.e., certain toxicities such as alopecia will not be considered in this category).
10. Ability to comply with study procedures, including hospitalization and protocol-specified acquisition of blood and/or bone marrow specimens.
11. Willing to be followed up long term, i.e. a 15-year follow up as required by health authorities for cell and gene therapy products.
12. Women of childbearing potential must test negative for pregnancy at enrolment and during the study.

Exclusion Criteria:

At screening: patients must meet none of the following exclusion criteria to be eligible for the study:

1. History of or candidate for allogeneic stem cell transplantation.
2. Cardiovascular, pulmonary, renal, and hepatic functions that in the judgment of the investigator are insufficient for the patient to undergo investigational CAR T-cell therapy.
3. Any history of or suspected current autoimmune disorders (apart from vitiligo, resolved childhood atopic dermatitis, Graves' disease clinically controlled).
4. History of rheumatologic disorders requiring specific treatment at any time in the patient's medical history.

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Ciceri, MD, Principal Investigator — IRCCS San Raffaele
Locations (3):
- Department of Haematooncology, Fakultni Nemocnice, Ostrava, Czech Republic, Czechia
- Italy (2):
  - IRCCS San Raffaele, Milan
  - IRCCS Ospedale Pediatrico Bambino Gesù, Roma

REFERENCES:
- [Derived] Stornaiuolo A, Valentinis B, Sirini C, Scavullo C, Asperti C, Zhou D, Martinez De La Torre Y, Corna S, Casucci M, Porcellini S, Traversari C. Characterization and Functional Analysis of CD44v6.CAR T Cells Endowed with a New Low-Affinity Nerve Growth Factor Receptor-Based Spacer. Hum Gene Ther. 2021 Jul;32(13-14):744-760. doi: 10.1089/hum.2020.216. Epub 2021 May 5. PMID 33554732

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population originally planned is made up of: Adult patients 18 to 75 years old or 18 to 63 years old for CZ site, with relapsed/refractory AML or MM expressing CD44v6; Children 1 to 17 years old with AML, only in Phase IIa, except for CZ site. Up to the early termination of the study only adult patients 18 to 75 years old or 18 to 63 years old for CZ site, with relapsed/refractory MM expressing CD44v6 were recruited
Pre-assignment Details: The recruited patient population, due to the early termination of the clinical study, was made up only of patients affected by multiple myeloma (MM), whereas AML patients were not enrolled.
  Eight patients, 6 males and 2 females were enrolled in 2 centers. Two patients received the investigational product (MLM-CAR44.1 T-cells), while 6 patients did not. Age ranged from 41 to 66 years, with a median of 56 years.
Groups:
- MLM-CAR44.1 T-cells Infusion: Patients were scheduled to receive a single intravenous (iv) infusion of CD44v6.CAR-transduced autologous lymphocytes at day 0, after lymphodepleting chemotherapy with cyclophosphamide iv (500 mg/m2) and fludarabine iv (30 mg/m2) performed daily from day -5 to day -3
  The dose of iv infused MLM-CAR44.1 T-cells is:
  PHASE I: 0.5x10E6/Kg or 1x10E6/Kg or 2x10E6/Kg according to the BOIN design. PHASE IIa: a dose of MLM-CAR44.1 T-cells corresponding to the maximum tolerated dose (MTD).
Period: Overall Study
Arm/Group | MLM-CAR44.1 T-cells Infusion
Started | 8 (Enrolled patients. Overall, 8 patients were enrolled in the study and underwent the screening phase to evaluate the compliance to the clinical inclusion / exclusion criteria as well as the CD44v6 expression by tumor cells.)
Treated Patients | 2 (Of the 8 enrolled patients, 2 were treated with MLM-CAR44.1 T-cell at the first dose level.)
Completed | 1
Not Completed | 7
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1
Not completed — Screening Failure | 5

BASELINE CHARACTERISTICS:
Population: Overall, 8 patients were enrolled in the study and underwent the screening phase to evaluate the compliance to the clinical inclusion / exclusion criteria as well as the CD44v6 expression by tumor cells (Table 10).
  Of the 8 enrolled patients, 2 were treated with MLM-CAR44.1 T-cell at the first dose level. Five patients were screening failures and 1 patient dropped-out before lymphocyte apheresis for fulminant disease progression.
Arm/Group | MLM-CAR44.1 T-cells Infusion
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 56 [41 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Italy | 5
  Czechia | 3
Confirmed diagnosis of MM [Count of Participants; unit: Participants] | 8
Patients with relapse or refractory disease [Count of Participants; unit: Participants] | 8

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Maximum Tolerated Dose (MTD) and the Recommended Phase IIa Dose of MLM-CAR44.1 T-cells in AML and MM
Description: MTD established through BOIN design and the dose-limiting toxicities (DLTs) occurring following CAR T-cell infusion.
Time Frame: Within 30 days following CAR T-cell infusion, assessed as day 0
Population: Data were not collected due to early end of trial
Arm/Group | MLM-CAR44.1 T-cells Infusion
Number analyzed (Participants) | 0

2. Primary Outcome: Phase I: Overall Safety of Treatment With MLM-CAR44.1 T-cells
Description: Safety will be evaluated by analyzing the type, frequency and severity of adverse events (AE) and by monitoring for systemic reactions (fever, tachycardia, nausea and vomiting, joint pain, skin rash).
  Overall, 3 study emergent serious adverse events (SAEs) were reported in patients treated with MLM-CAR44.1 T-cells.
Time Frame: For 30 days following CAR T-cell infusion, assessed as day 0.
Measure: Number; unit: Number of SAEs
Arm/Group | MLM-CAR44.1 T-cells Infusion
Number analyzed (Participants) | 2
Number of SAEs | 3

3. Primary Outcome: Phase I: Absence of Replication Competent Retrovirus (RCR) in Blood Specimens: 3 Months Post-infusion
Description: The absence of replication competent retrovirus (RCR) in blood specimens: 3 months post-infusion will be monitored by DNA PCR for the Galv gene.
  RCR search was conducted centrally using a quantitative molecular test, (real time quantitative PCR, q-PCR analysis) determining the absence of RCR by DNA PCR for the Galv and gag-pol genes on genomic DNA from patient's peripheral blood lymphocytes. The objective of this q-PCR analysis is to exclude the presence of RCR originated by recombination with PG13 packaging cell sequences by detecting the Galv and gag-pol transcripts in the transduced cells. The absence of the Galv and gag-pol transcripts can exclude the presence of an RCR, while its presence is not sufficient to indicate the presence of an RCR, and in this case further analysis is required.
Time Frame: 3 months after infusion (assessed as day 0)
Measure: Count of Participants; unit: Participants
Arm/Group | MLM-CAR44.1 T-cells Infusion
Number analyzed (Participants) | 2
Participants | 2

4. Primary Outcome: Phase I: Absence of Replication Competent Retrovirus (RCR) in Blood Specimens: 6 Months Post-infusion
Description: The absence of replication competent retrovirus (RCR) in blood specimens will be monitored by DNA PCR for the Galv gene.
  RCR search was conducted centrally using a quantitative molecular test, (real time quantitative PCR, q-PCR analysis) determining the absence of RCR by DNA PCR for the Galv and gag-pol genes on genomic DNA from patient's peripheral blood lymphocytes. The objective of this q-PCR analysis is to exclude the presence of RCR originated by recombination with PG13 packaging cell sequences by detecting the Galv and gag-pol transcripts in the transduced cells. The absence of the Galv and gag-pol transcripts can exclude the presence of an RCR, while its presence is not sufficient to indicate the presence of an RCR, and in this case further analysis is required
Time Frame: 6 months after infusion (assessed as day 0)
Measure: Count of Participants; unit: Participants
Arm/Group | MLM-CAR44.1 T-cells Infusion
Number analyzed (Participants) | 2
Participants | 2

5. Primary Outcome: Phase I: Absence of Replication Competent Retrovirus (RCR) in Blood Specimens: 12 Months Post-infusion
Description: The absence of replication competent retrovirus (RCR) in blood specimens will be monitored by DNA PCR for the Galv gene.
Time Frame: 12 months after infusion (assessed as day 0)
Population: Data were not collected due to early end of trial
Arm/Group | MLM-CAR44.1 T-cells Infusion
Number analyzed (Participants) | 0

6. Primary Outcome: Phase I: Absence of Replication Competent Retrovirus (RCR) in Blood Specimens: 24 Months Post-infusion
Description: The absence of replication competent retrovirus (RCR) in blood specimens will be monitored by DNA PCR for the Galv gene.
Time Frame: 24 months after infusion (assessed as day 0)
Population: Data were not collected due to early end of trial
Arm/Group | MLM-CAR44.1 T-cells Infusion
Number analyzed (Participants) | 0

7. Primary Outcome: Phase IIa: Hematological Disease Response to MLM-CAR44.1 T-cells in AML.
Description: The hematologic disease response will be classified according to ELN criteria.
Time Frame: 2 months after MLM-CAR44.1 T-cell infusion, assessed as day 0
Population: Data were not collected because Phase IIa was not performed due to early end of trial
Arm/Group | MLM-CAR44.1 T-cells Infusion
Number analyzed (Participants) | 0

8. Primary Outcome: Phase IIa: Hematological Disease Response to MLM-CAR44.1 T-cells in MM
Description: The hematologic disease response will be classified according to IMWG criteria
Time Frame: 3 months after T-cell infusion, assessed as day 0
Population: Data were not collected because Phase IIa was not performed due to early end of trial
Measure: Count of Participants; unit: Participants
Arm/Group | MLM-CAR44.1 T-cells Infusion
Number analyzed (Participants) | 2
Participants | 0

9. Secondary Outcome: Phase I: Hematologic Disease Response to MLM-CAR44.1 T-cells in AML
Description: The hematologic disease response will be classified with the following response criteria: complete response (CR), incomplete response (CRi) and partial response (PR) according to ELN criteria.
Time Frame: 1 and 2 months following T-cell infusion, assessed as day 0
Population: Data were not collected because no AML patients were enrolled
Arm/Group | MLM-CAR44.1 T-cells Infusion
Number analyzed (Participants) | 0

10. Secondary Outcome: Phase I: Hematologic Disease Response to MLM-CAR44.1 T-cells in MM
Description: Hematologic disease response evaluated at Day 28 following CART-cell infusion, as overall response rate (ORR), stringent complete response (sCR), CR, very good partial response (VGPR) and partial response (PR).
Time Frame: 1 and 3 months following T-cell infusion, assessed as day 0
Population: Hematologic disease response of the two treated patients was evaluated at Day 28 following CART-cell infusion. Both patients showed a progressive disease (PD) and no sign of response.
Measure: Count of Participants; unit: Participants
Arm/Group | MLM-CAR44.1 T-cells Infusion
Number analyzed (Participants) | 2
Participants
  No response detected | 2
  Hematologic disease response | 0

11. Secondary Outcome: Phase I: The Levels of Circulating MLM-CAR44.1 T-cells in Blood Samples
Description: The levels will be evaluated by flow cytometry and qPCR (in vivo pharmacokinetic profile).
Time Frame: At day 7, 14, 21, 28, 60, 90, 180 from infusion, assessed as day 0
Measure: Count of Participants; unit: Participants
Arm/Group | MLM-CAR44.1 T-cells Infusion
Number analyzed (Participants) | 2
Participants
  Positive at day 14 and 21 | 1
  Negative at all monitoring time points | 1

12. Secondary Outcome: Phase I: The Percentage of Patients for Whom Activation of Suicide Gene Was Needed
Description: Suicide gene activation and elimination of transduced cells will be established through administration of ganciclovir in case of cytokine-release syndrome (CRS) and other MLM-CAR44.1 T-cell related toxicities.
Time Frame: At day 7, 14, 21, 28, 60, 90, 180 from infusion, assessed as day 0
Population: Data were not collected because no MLM-CAR44.1 T-cell related toxicities occurred
Groups:
- MLM-CAR44.1 T-cells Infusion: Patients were scheduled to receive a single intravenous (iv) infusion of CD44v6.CAR-transduced autologous lymphocytes at day 0, after lymphodepleting chemotherapy with cyclophosphamide iv (500 mg/m2) and fludarabine iv (30 mg/m2) performed daily from day -5 to day -3
  The dose of iv infused MLM-CAR44.1 T-cells is:
  PHASE I: 0.5x10E6/Kg or 1x10E6/Kg or 2x10E6/Kg according to the BOIN design.
Arm/Group | MLM-CAR44.1 T-cells Infusion
Number analyzed (Participants) | 0

13. Secondary Outcome: Phase IIa: Hematologic Disease Response in AML
Description: as for outcome 9
Time Frame: 1, 2 and 6 months after MLM-CAR44.1 T-cell infusion, assessed as day 0.
Population: Data were not collected because Phase IIa was not performed due to early end of trial
Arm/Group | MLM-CAR44.1 T-cells Infusion
Number analyzed (Participants) | 0

14. Secondary Outcome: Phase IIa: Hematologic Disease Response in MM
Description: The hematologic disease response will be defined based on the overall response rate (ORR): stringent complete response (sCR), complete response (CR), very good partial response (VGPR), and partial response (PR) according to IMWG criteria
Time Frame: 1, 2 and 6 months after T-cell infusion, assessed as day 0
Population: Data were not collected because Phase IIa was not performed due to early end of trial
Arm/Group | MLM-CAR44.1 T-cells Infusion
Number analyzed (Participants) | 0

15. Secondary Outcome: Phase IIa: Overall Survival (OS)
Description: Overall Survival (OS) is defined as the time from the date of MLM-CAR44.1 T-cell infusion to the date of last follow-up or death due to any cause, whichever occurs first. One patients out of the 2 treated was still alive at the date of the early study termination. One patient died after EURE-CART-1 cell infusion, at day 121, for disease progression.
Time Frame: At the date of the early study termination
Population: Data were not collected because Phase IIa was not performed due to early end of trial
Arm/Group | MLM-CAR44.1 T-cells Infusion
Number analyzed (Participants) | 0

16. Other Pre Specified Outcome: Exploratory Outcome of Phase IIa: Percentages of Patients With Minimal Residual Disease
Description: AML: proportion of patients with a molecular complete response (CR); MM: proportion of patients with a molecular CR.
Time Frame: AML: 2 months after infusion, assessed as day 0. MM: 3 months after infusion, assessed as day 0
Population: Data were not collected because Phase IIa was not performed due to early end of trial
Arm/Group | MLM-CAR44.1 T-cells Infusion
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 15 months
Description: All SAEs and AEs are collected regardless of their relationship with the experimental product. Laboratory abnormalities that constitute an AE should be recorded on the Adverse Events page of the eCRF. Whenever possible, a diagnosis, rather than a symptom should be provided. Laboratory abnormalities that meet the criteria for Adverse Events should be followed until they have returned to normal or an adequate explanation of the abnormality is found.
Arm/Group | MLM-CAR44.1 T-cells Infusion
All-Cause Mortality (participants affected / at risk) | 1/2
Serious Adverse Events (participants affected / at risk) | 2/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MLM-CAR44.1 T-cells Infusion (N=2)
Pneumonia (Infections and infestations) | 2
Disease progression (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MLM-CAR44.1 T-cells Infusion (N=2)
Pyrexia (Immune system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 2
Anemia (Blood and lymphatic system disorders) | 2

LIMITATIONS AND CAVEATS:
The early termination of this study is due to the analysis of its feasibility, based on the low patient recruitment rate (due to the lower-than-expected proportion of myeloma and leukemia expressing the CD44v6). A further decrease in the recruitment occurred with the diffusion of the COVID-19 emergency and the availability of new drugs for the treatment of myeloma and leukemia. These reasons make impossible to foresee the conclusion of the study in a clinically relevant time frame.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Company will keep the information related to the trial in the strictest confidence and won't disclose such confidential information to third parties without the written consent of the Sponsor. It warrants that the obligation of confidentiality will be extended to the PI, his collaborators and to any other person who may become aware of confidential data. These obligations will remain in effect until the information is released into the public domain by the by the Sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-08): https://cdn.clinicaltrials.gov/large-docs/01/NCT04097301/Prot_SAP_000.pdf